CLINICAL TRIAL: NCT05774015
Title: The Effect of Oral Magnesium Supplementation on The Control and Outcomes of Type II Diabetes Mellitus Guided by Serum Ionized Magnesium Level: A Double-Blind Randomized Control Trial
Brief Title: Effect of Oral Magnesium Supplementation on Type II Diabetes Mellitus Guided by Serum Ionized Magnesium Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Qaboos University (Other)
Collaborators: Nova Biomedical (Industry)
Responsible Party: Principal Investigator, Prof. Mohammed Al za'abi, Professor, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SQUH-ionized magnesium
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes; Magnesium Disorder
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Magnesium Oxide

STUDY DESIGN:
Intervention Model Description: A prospective double-blind RCT with a control group and an interventional group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Mg oxide tablets or placebo tablets (a total of 4 bottles, 90 tablets in each coded bottle) will be provided for each participant during the study period. The 4 bottles for each participant will be per-coded to match the randomization labels to ensure a double-blinded process
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group (Mg oxide supplementation): (Active Comparator): Interventional group (Mg oxide supplementation): Patients in this group will receive Mg oxide tablet 500 mg (302 mg elemental), with a dosage regimen of 1 table once daily as per the recommended range of the daily dose (from 250 to 500 mg elemental) (29, 31, 41, 45). Tablets should be taken with food and 2 hrs. apart from other medications for 12 consecutive months.
  Interventions: Dietary Supplement: Magnesium Oxide tablet 500 mg
- Control group (placebo tablets) (Placebo Comparator): Control group (placebo tablets): Patients in this group will receive placebo tablets labeled as 500 mg (302 mg elemental), with a dosage regimen of 1 tablet once daily. Tablets should be taken with food and 2 hrs. apart from other medications for 12 consecutive months.
  Interventions: Dietary Supplement: Magnesium Oxide tablet 500 mg

INTERVENTIONS:
Dietary Supplement: Magnesium Oxide tablet 500 mg — To supplement T2DM with Mg oxide tablets (500 mg total, 302 mg elemental) regardless on their magnesium level

SUMMARY:
Studies have shown that type 2 diabetic patients (T2DM) may have low serum magnesium levels leading to poor control and outcome of the disease. Supplementation with Mg might improve overall diabetic control and disease outcome. However, there is yet no consensus on whether the ionized (iMg) or the total Mg (tMg) level should be used as a basis to determine the status of Mg in the blood. Recently it was shown that iMg may correlate better with diabetes control than tMg. Therefore, Mg supplements to diabetic patients may improve their disease status. Unfortunately, and to the best of our knowledge all of the available trials on Mg supplementation guided by iMg levels were conducted on healthy volunteers rather than T2DM patients, and they were all for a short period of time (10 days to 10 weeks). Here we hypothesize that supplementations of T2DM patients with Mg based on serum iMg levels correlate better with diabetes control and prognosis. Such hypothesis is supported by a retrospective study that concluded that iMg correlate better with BP control than tMg. In addition, another trial that investigated the effects of three Mg dietary supplements; Mg oxide, Mg citrate and Mg carbonate on healthy female young adults, showed that only Mg oxide led to an increase in the levels of iMg and tMg concentrations when compared to baseline. Furthermore, a case-control study on older diabetic patients revealed a significant association between iMg and HbA1c. This study aims to investigate the effect of supplementing Mg oxide tablets versus placebo tablets guided by serum iMg levels in T2DM patients with or without hypomagnesemia on diabetic control and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old).
* Treated with oral hypoglycemic agents (OHA) ± insulin regimen.
* Had HbA1c ≥ 7% in the last 3 months

Exclusion Criteria:

* HbA1c of < 7%.
* Fully dependent patients as per clinical frailty score
* End stage renal disease (creatinine clearances (CrCl) at < 10ml/min)
* With neuromuscular disease
* With active solid or hematological malignancies.
* With cognitive disorders.
* With the following regular medications (baloxavir marboxil, calcium/sodium polystyrene sulfate, raltegravir, or unithiol) due to X category drug-drug interaction (contraindicated combinations) when given concurrently Mg oxide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c%) | 3-month and 12-month
  To evaluate the reduction in HbA1c% levels after 3 and 12 months of Mg supplementation versus placebo between the interventional group verse the control group.
Fasting Blood Glucose (FBG) | 3-month and 12-month
  To evaluate the reduction in FBG levels after 3 and 12 months of Mg supplementation versus placebo between the interventional group verse the control group.

SECONDARY OUTCOMES:
Emergency department (ED) visits, hospital admission, and length of hospital stay (LOS) | 3-month and 12-month
  To determine the rate of ED visits, hospital admission, and LOS after 3 months and 12 months of Mg supplementation between the interventional group verse the control group.
Total dosage of insulin regimen | 3-month and 12-month
  To evaluate the pattern of total dosage adjustment in the insulin regimen after 3 months and 12 months of Mg supplementation versus placebo between the interventional group verse the control group.
Blood pressure | 3-month and 12-month
  To evaluate the reduction BP measurement after 3 months and 12 months of Mg supplementation versus placebo between the interventional group verse the control group.
lipid profile | 3-month and 12-month
  To evaluate the reduction in lipid profile after 3 and 12 months of Mg supplementation versus placebo between the interventional group verse the control group.
Serum creatinine | 3-month and 12-month
  To evaluate the rate of changes in serum creatinine after 3 and 12 months of Mg supplementation versus placebo between the interventional group verse the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammed AlZa'abi, Muscat, Oman

IPD SHARING:
Plan to Share IPD: Yes
the whole IPD can be shared
Supporting Information: Study Protocol
Time Frame: no limits